CLINICAL TRIAL: NCT06032390
Title: Artificial Intelligence in BreastScreen Norway - a Randomized Controlled Trial
Brief Title: Artificial Intelligence in Mammography Screening in Norway
Acronym: AIMS Norway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Helse Vest (Other); Helse Midt-Norge (Other); Helse Nord (Industry); Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 366405
Record Dates: First submitted 2023-07-05; First posted 2023-09-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Screening; Digital Mammography; Artificial Intelligence; Randomized Controlled Trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to an intervention or control arm. Intervention arm will be triaged based on AI result score.
Who Masked: Participant, Care Provider
Masking Description: Neither the participant nor the radiologic technician performing the mammography examination will know to what study arm the participant was allocated. Radiologists reading the screening examinations will be blinded to the intervention at initial reading but not in the consensus meeting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): AI assisted mammography screening interpretation
  Interventions: Other: AI assisted mammography screening interpretation
- Control arm (Active Comparator): Standard mammography screening interpretation (standard procedure)
  Interventions: Other: Standard mammography screening interpretation

INTERVENTIONS:
Other: AI assisted mammography screening interpretation — Screening examinations will be analyzed by the AI system (Transpara, ScreenPoint Medical, Nijmegen, The Netherlands) that assigns each examination a cancer risk score 1-10. Examinations with a score 1-7 will be single read and examinations with score 8-10 will be double read. Examinations selected by one or two readers will be discussed in a consensus meeting. Examinations with an AI score of >9.8 will be selected for the consensus meeting by default. AI risk scores and image markings are provided to the readers only in the consensus meetings. The readers will decide whether to recall the woman for further assessment in consensus (standard procedure).
  Arms: Intervention arm
Other: Standard mammography screening interpretation — Screening examinations will be assessed according to standard of care: independently double read, examinations selected by one or two readers will be discussed in a consensus meeting, and the radiologists will decide whether to recall the woman for further assessment. Screening examinations will be analyzed by the AI system retrospectively but the results will not be made available to the radiologist, only used for comparison to the intervention group in results analyses.
  Arms: Control arm

SUMMARY:
The purpose of this randomized controlled trial is to compare the number of breast cancers detected among women who had their screening mammograms interpreted by artificial intelligence (AI) in combination with one or two breast radiologists to the number of breast cancers detected after standard independent double reading in BreastScreen Norway. The aims of the study is to prove that screening interpretation with AI in combination with one or two radiologists (the intervention) is non-inferior to standard interpretation procedure.

DETAILED DESCRIPTION:
Independent double reading with consensus is the recommended practice for breast cancer screening programs in Europe. This is a time-consuming process and more than 99% of examinations are determined to have a negative final outcome in BreastScreen Norway. However, radiologist still overlook cancers, and review-studies have shown 20-25% of screen-detected and interval cancers to be visible at prior screening mammograms. In Norway and other countries, there is also a shortage of breast radiologists.

Retrospective studies on AI in mammographic screening have shown promising results in the classification of cancer negative and cancer positive examinations. However, prospective studies are needed to elucidate questions concerning AI as a support or replacement for the radiologists in the interpretation process.

In this randomized controlled trial women attending screening and consenting to participate in the study, will be randomized (1:1 allocation) to an intervention or a control group. The screening examination will be performed as usual in both groups. The intervention in the trial is the interpretation procedure.

All examinations will be analyzed by AI. In the intervention group, examinations will be triaged according to risk of malignancy defined by an AI score. Examinations with a low AI score (1-7) will have a single reading by one radiologist and examinations with a intermediate or high AI score (8-10) will have an independent double reading by two radiologists. All examinations selected by either one or both radiologist will be discussed at consensus. Examinations with an AI raw score of >9.8 will be discussed at consensus independent of the radiologists' interpretation. The radiologists will be blinded to whether the mammograms are interpreted by one or two radiologists. AI risk scores and AI image marking of suspicious calcifications and masses are only provided to the radiologists at consensus, not during independent reading. In the control group, two independent radiologists will interpret all screening examinations according to standard procedure, independent double reading. AI results will not be available at either independent reading or consensus, only for comparison with the intervention group in final analyses.

Screen-detected cancers in the intervention and control arm will be analyzed in terms of non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Women attending the population-based mammography screening program BreastScreen Norway providing a signed, informed consent

Exclusion Criteria:

* Women attending the population-based mammography screening program BreastScreen Norway not providing a signed, informed consent

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150000 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Screen-detected breast cancers | 36 months from study start-up
  Number of breast cancers detected at screening per 1000 screening examinations.

SECONDARY OUTCOMES:
Consensus rate | 24 months from study start-up
  Proportion of participant discussed in consensus among all participants (%).
Recall rate | 24 months from study start-up
  Proportion of women recalled for further assessment among all participants (%).
Interval breast cancers | 60 months from study start-up
  Number of interval breast cancers diagnosed per 1000 screening examinations.
Prognostic and predictive tumor characteristics of screen-detected breast cancer | 36 months from study start-up
  Distribution of tumor characteristics among the participants with screen-detected breast cancer.
Prognostic and predictive tumor characteristics of interval breast cancer | 60 months from study start-up
  Distribution of tumor characteristics among the participants with interval breast cancer.
Sensitivity | 60 months from study start-up
  Proportion of true positives among true positive and false negatives (%).
Specificity | 60 months from study start-up
  Proportion of true negatives among true negatives and false positives (%).
Mammographic features of screen-detected breast cancer | 36 months from study start-up
  Distribution of characteristics of tumors observed on the mammograms of participants diagnosed with screen-detected breast cancer.
Time spent screen-reading | 36 months from study start-up
  Time (minutes:seconds) spent by the individual radiologists interpreting screening mammograms

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Hofvind, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Cancer Registry of Norway, Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside the project group.